CLINICAL TRIAL: NCT05939011
Title: Pilot Investigation of the Ketogenic Diet's Health Effects Through Multi-Omics Assessment
Brief Title: Ketogenic Diet Health and Longevity
Acronym: KDHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Debra K. Sullivan, PhD, RD, Department Chair, Dietetics and Nutrition, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY147643
Record Dates: First submitted 2023-02-10; First posted 2023-07-11 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Ketogenic Dieting; Ketoses, Metabolic; Ketosis
Keywords: ketogenic; well-formulated ketogenic diet; keto
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Single-arm, pilot clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Well-formulated ketogenic diet (WFKD) (Experimental): The researchers aim to enroll 20 healthy adults recruited from Kansas City and surrounding areas for an 8-week WFKD diet intervention. Study personnel will obtain baseline (week 0), mid-point (week 4), and end-of-study (8 weeks) blood samples, anthropometrics, and dietary intake data. Fecal microbiome samples and dual energy x-ray absorptiometry (DXA) are collected at baseline and 8-weeks. Blood samples collected at baseline and 8-week visits will be measured for metabolic biomarkers, inflammatory biomarkers, and RNA. The blood sample collected at the 4-week visit will include glucose, insulin, insulin resistance, and beta-hydroxybutyrate to track diet adherence and adjust the diet as needed.
  Interventions: Behavioral: Well-formulated Ketogenic Diet

INTERVENTIONS:
Behavioral: Well-formulated Ketogenic Diet — 1:1 ketogenic diet that is focused on intake of high-quality fats (nuts/seeds, fatty fish, avocado) and reduction in processed food.

SUMMARY:
The goal of this pilot intervention is to learn about how a well-formulated ketogenic diet (WFKD) impacts various health factors in generally healthy adults. The main questions it aims to answer are:

* Establish whether an 8-week isocaloric, WFKD improves body composition and metabolic biomarkers in adults without chronic disease.
* Examine changes in transcriptomic sequencing pathways pre- and post-WFKD intervention.
* Explore gut microbial changes in adults without chronic disease that consume a WFKD.

Participants will follow a well-formulated ketogenic diet for 8-weeks. Study procedures include:

* Weekly body weight tracking
* Daily urinary ketone assessment
* Pre/post stool samples for gut microbiota analyses
* Pre/post DXA scans
* Diet quality tracking through 3-day food records

ELIGIBILITY:
Inclusion Criteria:

* 30 to 55 years
* Speaks English as primary language
* BMI 20.0-34.9 kg/m^2

Exclusion Criteria:

* Certain medications (statin, blood pressure, thyroid hormone replacement, etc.)
* Prior medical diagnosis of type 1 or type 2 diabetes mellitus, cancer requiring chemotherapy or radiation therapy within 5 years, cardiac event, GI disorders, traumatic brain injury/multiple concussions, hypertension, dyslipidemia, or any diagnosis deemed ineligible by study team
* History of renal stones
* Currently lactating
* Already following a ketogenic diet
* Adherence to a specialized diet regimen that disallows compliance
* Use of tobacco or tobacco replacement products within 1 year

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in Body Composition-- dual x-ray absorptiometry (DXA) | Baseline, 8 Week
  Measures of tissue distribution
Changes in Waist Circumference (WC) | Baseline, 4 Week, 8 Week
  Waist circumference (cm)
Changes in Body Mass Index (BMI) | Baseline, 4 Week, 8 Week
  Ratio of height and weight in kg/m^2
Changes in Homeostatic model assessment of Insulin Resistance (HOMA-IR) | Baseline, 4 Week, 8 Week
  Ratio of fasting glucose and fasting insulin with a conversion factor, unitless
Changes in Advanced Lipid Panel | Baseline, 8 Week
Changes in Inflammation | Baseline, 8 Week
  Changes in high sensitivity C-reactive protein (hs-CRP) (mg/L)

SECONDARY OUTCOMES:
Changes in transcriptomic sequencing pathways | Baseline, 8 weeks
  Measured via RNASequencing (RNA-Seq) technique: high-throughput (~25,000 genes) RNAseq using SE100 Illumina (HiSeq) reads
Gut microbial changes | Baseline, 8 weeks
  Taxonomic classification of individual operational taxonomic units (OTU) with 97% similarity and produce an OTU table of all identified taxa across all samples

CONTACTS AND LOCATIONS:
Overall Officials: Debra K Sullivan, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No